CLINICAL TRIAL: NCT07345845
Title: Contribution of Mineralocorticoid Receptor Signaling to Vascular Dysfunction & Aberrant Inflammation After Preeclampsia
Brief Title: MR and Inflammation After Preeclampsia
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anna Stanhewicz, PhD (Other)
Responsible Party: Sponsor-Investigator, Anna Stanhewicz, PhD, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202508378
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Preeclampsia; Preeclampsia Postpartum
MeSH Terms: conditions — Pre-Eclampsia | interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Assessment of microvascular function (Experimental): The investigators use intradermal microdialysis to deliver eplerenone and L-NAME to the cutaneous microvasculature
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — Local heating: eplerenone is locally and acutely delivered to the cutaneous microvasculature during local heating of the skin to assess endothelium-dependent dilation, L-NAME is added to assess nitric oxide-dependent dilation during this response

SUMMARY:
The purpose of this investigation is to examine the role of inappropriate mineralocorticoid receptor activation in endothelial dysfunction and vascular inflammation in otherwise healthy women with a history of preeclampsia. The main questions it aims to answer are:

1. Does overactivation of the mineralocorticoid receptor contribute to reduced endothelial function in women who had preeclampsia?
2. To what extent does the mineralocorticoid receptor mediated exaggerated production of inflammatory cytokines in immune cells from women who had preeclampsia?

Participants will visit the research laboratory for 2 experimental visits:

* Visit 1: Skin blood flow will be measured using a minimally invasive technique (intradermal microdialysis for the local delivery of pharmaceutical agents) to examine blood vessels in a nickel-sized area of the skin.
* Visit 2: Endothelial cells will be collected from an antecubital vein.

ELIGIBILITY:
Inclusion Criteria:

* women who had preeclampsia and women who did not have preeclampsia
* 12 weeks to 5 years postpartum
* 18-45 years old

Exclusion Criteria:

* history of hypertension or metabolic disease before pregnancy
* history of gestational diabetes
* history of gestational hypertension without preeclampsia
* skin diseases
* current tobacco use
* current antihypertensive medication
* statin or other cholesterol-lowering medication
* currently pregnant
* body mass index less than 18.5 kg/m2
* allergy to materials used during the experiment.(e.g. latex),
* known allergy to study drugs or salt-supplement

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in microvascular endothelial function following local eplerenone treatment compared to placebo treatment measured by laser-Doppler flowmetry | post 1 hour of skin perfusion
  Cutaneous vascular vasodilator response (cutaneous conductance; %max) to local heating of the skin; intradermal microdialysis for the local delivery of eplerenone compared to control (Ringer's solution), followed by L-NAME infusion to quantify NO-dependent response

SECONDARY OUTCOMES:
Mineralocorticoid receptor expression in endothelial cells | a total of 1 time during the study, within ~4 weeks following enrollment
  The investigators will quantify expression of the mineralocorticoid receptor in biopsied endothelial cells.
Inflammatory response from isolated immune cells | from a blood draw collected at the start of the experimental visit
  The investigators will measure inflammatory responses, assessed as inflammatory cytokine release following activation of immune cells in the presence and absence of eplerenone treatment. Cells are collected from a blood draw and treated with eplerenone in a cell culture environment (ex vivo treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Reid-Stanhewicz, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No